CLINICAL TRIAL: NCT06289335
Title: Dexmedetomidine Compared With Ondansetron in Treating Postanesthetic Shivering in Patients After Regional Anesthesia for Cesarean Section-a Randomized Clinical Trial.
Brief Title: Dexmedetomidine Compared to Ondansetron for Postanaesthetic Shivering in Patients Undergoing a Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, MARIO AURELIO MARTÍNEZ-JIMÉNEZ, Doctor, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCDrIMPrieto anaesthesia
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Postanesthetic Excitement; Cesarean Section
Keywords: shivering, dexmedetomidine, ondansetron, regional anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Saline Solution; Isotonic Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): 0.3 mcg Kg-1 (actual weight) of dexmedetomidine IV in 20 mL of saline
  Interventions: Drug: saline solution
- Ondansetron (Sham Comparator): 8 mg ondansetron IV in 20 mL saline
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: saline solution — 20 mL of saline
  Other Names: isotonic solution

SUMMARY:
Evaluate the efficiency of management with intravenous dexmedetomidine compared to intravenous ondansetron to achieve the disappearance of post-anesthetic shivering in a shorter time in the obstetric patient undergoing cesarean section under regional anesthesia.

DETAILED DESCRIPTION:
Randomized clinical trial with 40 pregnant patients, between 18 and 45 years old with ASA (American Society of Anesthesiologist) II or III, undergoing scheduled or emergency cesarean section with regional anesthesia and who presented grade tremor 1 based on the BSAS (Bedside shivering assessment scale) scale, at the Hospital Central from San Luis Potosi, Mexico. The main objective of this study was to quantify the time that elapsed from the end of the administration of the medication until the disappearance of the tremor, which was measured in minutes; The evaluation of the disappearance, persistence or reappearance of the tremor was solely visual by the anesthesiology staff.

ELIGIBILITY:
Inclusion Criteria:

* ASA II or III, undergoing scheduled or emergency cesarean section with regional anesthesia (hyperbaric bupivacaine 0.5% with morphine at 1 mcg Kg-1) and who presented tremor grade >1 based on the BSAS scale

Exclusion Criteria:

* Hemodynamic instability, heart disease or sinus bradycardia, allergy to any of the medications applied, psychiatric diseases or hypothermia <35.2 ºC measured by tympanic temperature.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Period of time | one hour
  period of time in which post-anesthetic tremor is controlled from the moment of administration

SECONDARY OUTCOMES:
Adverse effects | one hour
  To measure the frequencies of occurrence of adverse effects and changes in vital signs (heart rate, blood pressure, and temperature [measured at the tympanic membrane]) correlated with resolution of tremor.

CONTACTS AND LOCATIONS:
Overall Officials: MARIO A MARTÍNEZ-JIMÉNEZ, Dr., Study Director — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No
It might be useful for other researchers to expand their investigations, nevertheless, in this moment it seems completed this branch of investigation.

REFERENCES:
- [Background] Lopez MB. Postanaesthetic shivering - from pathophysiology to prevention. Rom J Anaesth Intensive Care. 2018 Apr;25(1):73-81. doi: 10.21454/rjaic.7518.251.xum. PMID 29756066
- [Background] Jain A, Gray M, Slisz S, Haymore J, Badjatia N, Kulstad E. Shivering Treatments for Targeted Temperature Management: A Review. J Neurosci Nurs. 2018 Apr;50(2):63-67. doi: 10.1097/JNN.0000000000000340. PMID 29278601
- [Background] Tsai YC, Chu KS. A comparison of tramadol, amitriptyline, and meperidine for postepidural anesthetic shivering in parturients. Anesth Analg. 2001 Nov;93(5):1288-92. doi: 10.1097/00000539-200111000-00052. PMID 11682416
- [Background] Talke P, Tayefeh F, Sessler DI, Jeffrey R, Noursalehi M, Richardson C. Dexmedetomidine does not alter the sweating threshold, but comparably and linearly decreases the vasoconstriction and shivering thresholds. Anesthesiology. 1997 Oct;87(4):835-41. doi: 10.1097/00000542-199710000-00017. PMID 9357885
- [Background] Elvan EG, Oc B, Uzun S, Karabulut E, Coskun F, Aypar U. Dexmedetomidine and postoperative shivering in patients undergoing elective abdominal hysterectomy. Eur J Anaesthesiol. 2008 May;25(5):357-64. doi: 10.1017/S0265021507003110. Epub 2008 Jan 21. PMID 18205960
- [Result] Hoffman J, Hamner C. Effectiveness of dexmedetomidine use in general anesthesia to prevent postoperative shivering: a systematic review. JBI Database System Rev Implement Rep. 2016 Jan 15;13(12):287-313. doi: 10.11124/jbisrir-2015-2257. PMID 26767820
- [Result] Yu G, Jin S, Chen J, Yao W, Song X. The effects of novel alpha2-adrenoreceptor agonist dexmedetomidine on shivering in patients underwent caesarean section. Biosci Rep. 2019 Feb 1;39(2):BSR20181847. doi: 10.1042/BSR20181847. Print 2019 Feb 28. PMID 30643009
- [Result] Abdel-Ghaffar HS, Mohamed SA, Fares KM, Osman MA. Safety and Efficacy of Dexmedetomidine in Treating Post Spinal Anesthesia Shivering: A Randomized Clinically Controlled Dose-Finding Trial. Pain Physician. 2016 May;19(4):243-53. PMID 27228512
- [Result] He K, Zhao H, Zhou HC. Efficiency and safety of ondansetron in preventing postanaesthesia shivering. Ann R Coll Surg Engl. 2016 Jul;98(6):358-66. doi: 10.1308/rcsann.2016.0152. Epub 2016 May 3. PMID 27138855
- [Result] Nallam SR, Cherukuru K, Sateesh G. Efficacy of Intravenous Ondansetron for Prevention of Postspinal Shivering during Lower Segment Cesarean Section: A Double-Blinded Randomized Trial. Anesth Essays Res. 2017 Apr-Jun;11(2):508-513. doi: 10.4103/aer.AER_26_17. PMID 28663651
- [Result] Botros JM, Mahmoud AMS, Ragab SG, Ahmed MAA, Roushdy HMS, Yassin HM, Bolus ML, Goda AS. Comparative study between Dexmedetomidine and Ondansteron for prevention of post spinal shivering. A randomized controlled trial. BMC Anesthesiol. 2018 Nov 30;18(1):179. doi: 10.1186/s12871-018-0640-3. PMID 30501612